CLINICAL TRIAL: NCT00359255
Title: The Effect of a Supplementary Exercise Program for Upper Extremity Function in Stroke Rehabilitation
Brief Title: The Effect of Additional Arm Therapy on Arm Function After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Janice Eng, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: C05-0680; VO6-0117
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Stroke
Keywords: Exercise; rehabilitation; upper limb; inpatient; RCT; activities of daily living
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Behavioral: Education manual
- 2 (Experimental)
  Interventions: Behavioral: An inpatient homework based exercise program for the upper limb post stroke

INTERVENTIONS:
Behavioral: Education manual — The control arm was given education on stroke, the affected arm post strooke, bone health, and healthy living. This information was given in a booklet format and administered once weekly by the site coordinator.
  Arms: 1
Behavioral: An inpatient homework based exercise program for the upper limb post stroke — The experimental arm was given arm exercises graded based on motor impairment and administered by the site coordinator. The exercises were given in a booklet with written and photographic instructions. These exercises were monitored on a twice-weekly basis.
  The intervention was to be completed once daily for 45 minutes, 5 days per week, and supervised by the site coordinator. Exercises consisted of range of motion, strengthening, and use of the arm in daily activites such as buttoning, pouring and throwing.
  Arms: 2

SUMMARY:
This study would focus on a new method of adding extra arm exercise to the usual therapy delivered in the hospital. We propose to design an exercise program for the affected arm and hand that would be given to the client as homework and done in the client's hospital room. The program would be designed and monitored by a therapist that works in the hospital.

We believe that this program will: 1) increase arm and hand recovery over usual care received in the hospital, 2) help people make the move from therapist run exercise to self management of exercise, and 3) promote family involvement in therapy.

DETAILED DESCRIPTION:
In total 250 participants admitted for stroke rehabilitation at 4 BC sites will be randomly assigned to either the experimental or the control group. The extra arm and hand exercise program (experimental group) will receive usual therapy plus 60 minutes per day of additional arm exercises. This program will last for 4 weeks while the participant is in the hospital. The arm and hand program will include muscle strengthening and stretching, repetitive reaching, folding, stacking, pushing and pulling tasks, picking up objects, and activities that use speed and accuracy. The family will be encouraged to participate in the program with the participant. The control group will receive usual therapy only.

ELIGIBILITY:
Inclusion Criteria:

1. 19 years of age or older
2. arm recovery as a rehabilitation goal
3. have palpatable movement of wrist extension
4. able to follow 3 step verabal commands

Exclusion Criteria:

1. unstable cardiovascular status (congestive heart failure, uncontrolled hypertension, uncontrolled atrial fibrillation, or left ventricular failure),
2. significant musculo-skeletal problems (e.g., rheumatoid arthritis) or neurological conditions (e.g., Parkinson's disease) due to conditions other than stroke,
3. receptive aphasia

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the ability to use the paretic arm in activities of daily living. This outcome will be measured pre and post program.

SECONDARY OUTCOMES:
Secondary outcomes include amount of use and quality of movement of the paretic arm, motor recovery, strength, tone, and health related quality of life. Each of these measures will be evaluated pre and post program.

CONTACTS AND LOCATIONS:
Overall Officials: Janice Eng, Ph.D, Principal Investigator — The University of British Columbia
Locations (4):
- Canada (4):
  - Kelowna General Hospital, Kelowna, British Columbia
  - GF Strong Rehab Center, Vancouver, British Columbia
  - Holy Family Hospital, Vancouver, British Columbia
  - Victoria General Hospital, Victoria, British Columbia

REFERENCES:
- [Result] Harris JE, Eng JJ, Miller WC, Dawson AS. A self-administered Graded Repetitive Arm Supplementary Program (GRASP) improves arm function during inpatient stroke rehabilitation: a multi-site randomized controlled trial. Stroke. 2009 Jun;40(6):2123-8. doi: 10.1161/STROKEAHA.108.544585. Epub 2009 Apr 9. PMID 19359633